CLINICAL TRIAL: NCT03863535
Title: Panretinal Photocoagulation (PRP) vs PRP Combined With Intravitreous Conbercept (IVC) for Severe Nonproliferative Diabetic Retinopathy (nPDR): A Randomized Clinical Trial
Brief Title: PRP vs PRP+IVC for Severe nPDR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ruijin Hospital (Other)
Collaborators: Shanghai Municipal Science and Technology Commission (Other Government)
Responsible Party: Principal Investigator, Xi Shen, Department director of Ophthamology, Ruijin Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Ruijin Hospital
Record Dates: First submitted 2019-01-27; First posted 2019-03-05 (Actual); Last update posted 2019-03-05 (Actual); Status verified 2019-03

CONDITIONS: Severe Nonproliferative Diabetic Retinopathy; Diabetic Retinopathy; Diabete Mellitus
Keywords: Conbercept; Panretinal photocoagulation; non-proliferative diabetic retinopathy; diabetic macular edema
MeSH Terms: conditions — Diabetic Retinopathy; Diabetes Mellitus | interventions — KH902 fusion protein

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intravitreal conbercept+Panretinal coagulation (Experimental)
  Interventions: Drug: Conbercept; Procedure: Panretinal coagulation
- Panretinal coagulation (Active Comparator)
  Interventions: Procedure: Panretinal coagulation

INTERVENTIONS:
Drug: Conbercept — Participants were randomized (1:1) to receive IVC+PRP or PRP monotherapy. Patients in IVC+PRP group with diabetic macular edema (DME) received 3 monthly IVC injections along with standard PRP within 1 week after the first injection. Those without DME received 1 lVC injection and standard PRP within 1 week after the injection . Re-treatments in both groups were at the investigators'discretion.
  Arms: Intravitreal conbercept+Panretinal coagulation
Procedure: Panretinal coagulation — The PRP monotherapy group received standard PRP between day 1 and month 2; thereafter, re-treatments in both groups were at the investigators'discretion.

SUMMARY:
The randomized clinical trial aims to compare the therapeutic effects between panretinal photocoagulation(PRP) and PRP combined with intravitreal conbercept (IVC) injection in severe nPDR with/without diabetic macular edema patients.

DETAILED DESCRIPTION:
This was a prospective, randomized, two-armed study to assess the efficacy and safety of intravitreal conbercept injection plus PRP versus PRP in the treatment of nPDR patients with/without diabetic macular edema for a period of 1 year. This was an investigator-initiated study performed by department of ophthalmology, Ruijin hospital affiliated with Shanghai Jiaotong University School of Medicine.

ELIGIBILITY:
Inclusion Criteria:

Type II diabetic patients, 18 years and older, were included if the participants had:

1. severe non-PDR in either eyes with/without diabetic macular edema;
2. ETDRS letters-measured best-corrected visual acuity (BCVA) ranging from 20/40 to 20/320 Snellen equivalent;
3. no previous treatment (of any type) in either eye.

Exclusion Criteria:

1. history of prior laser treatment or vitrectomy in the study eye;
2. history of thromboembolic event - including myocardial infarction or cerebral vascular accident;
3. major surgery within the prior 6 months or planned within the next 28 days;
4. history of glaucoma or ocular hypertension;
5. loss of vision as a result of other causes;
6. history of systemic corticosteroid therapy within the last 3 months;
7. severe systemic disease other than diabetes mellitus;
8. known coagulation abnormalities or current use of anticoagulative medication other than aspirin
9. any condition that could affect followup or documentation (including preretinal or vitreous hemorrhage).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-01-18 (Actual); Primary Completion 2021-01-01 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in best-corrected visual acuity (BCVA) | from baseline to month 12
  To assess the effects of two therapies on visual acuity

SECONDARY OUTCOMES:
Change in central subfield thickness | from baseline to month 12
  optical coherence tomography (OCT) for the assessment of central macular thickness
Fundus fluorescein angiography | from baseline to month 12
  fluorescein angiography to measure area of fluorescein leakage (FLA)
Foveal avascular zone | from baseline to month 12
  Optical coherence tomography angiography (OCTA) for measurement of FAZ

CONTACTS AND LOCATIONS:
Overall Officials: Xi Shen, MD, Study Director — Ruijin Hospital; Qiong Zhang, MD, Principal Investigator — Ruijin Hospital
Locations (1):
- Ruijin Hospital, Shanghai, Shanghai Municipality, China